CLINICAL TRIAL: NCT05087654
Title: The Effects of a Combination of 3D Virtual Reality and Hands-on Horticultural Activities on Community-dwelling Older Adults' Mental Health: A Quasi-Experimental Study
Brief Title: 3D VR and Hands-on Horticultural Activities Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ECKIRB1090503
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Horticultural Therapy; Virtual Reality
Keywords: 3D virtual reality; horticultural therapy; community-dwelling; older adults; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Received the Combination of 3D VR and Hands-on Horticultural Activities.
  Interventions: Other: Combination of 3D VR and Hands-on Horticultural Activities
- Comparison group (No Intervention): Received scheduled activities, such as physical fitness, paper cutting, etc., without any gardening activities.

INTERVENTIONS:
Other: Combination of 3D VR and Hands-on Horticultural Activities — The intervention program consisted of 8 two-hour sessions that were conducted once a week for 8 consecutive weeks.
  Arms: Experimental group

SUMMARY:
This study aimed to explore the effects of a combination of 3D virtual reality (VR) and hands-on horticultural activities on the mental health of community-dwelling older adults.

DETAILED DESCRIPTION:
Aging societies are of public health concern worldwide. It is critical to develop strategies that harness technology to enhance older adults' mental health. This study aimed to explore the effects of a combination of three-dimensional virtual reality (3D VR) and hands-on horticultural activities on the mental health of community-dwelling older adults. Used a quasi-experimental design. A total of 62 community-dwelling older adults were recruited. The members of the experimental group participated in an 8-week intervention program. Participants of both groups completed before-and-after intervention measurements for outcome variables that included perceived self-esteem, depression, isolation, mastery and achievement motives, which were analyzed using the generalized estimating equation (GEE). This study found beneficial effects of a combination of 3D VR and hands-on horticultural activities on community-dwelling older adults' mental health.

ELIGIBILITY:
Inclusion Criteria:

Intact cognition, possessing the ability to understand verbal meaning and the ability to operate a VR joystick independently.

Exclusion Criteria:

A history of hand dysfunction, severe visual and hearing impairment, being allergic to plants or pollen, and a current illness such as epilepsy or stroke.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Self-esteem | about three months
  Rosenberg Self-Esteem Scale consists of 14 items and each item is scored on a Likert-type scale that ranges from 1 (strongly agree) to 4 (strongly disagree), with higher scores indicating a higher level of self-esteem.
Depression | about three months
  The Chinese version of the Geriatric Depression Scale was used, which has a total of 15 items. All items were answered as either yes (1) or no (0). The total raw scores ranged from 0 to 15, with a higher score indicating a higher level of depression.
Perceived isolation | about three months
  A short-form scale of perceived isolation was used to measure isolation. Each item was scored on a Likert-type scale from 1 (never) to 4 (often), with higher scores indicating a higher level of perceived isolation.
Perceived mastery | about three months
  The Chinese version of the Perceived Mastery Scale with a total of 7 items was used. Each item was scored on a Likert-type scale from 1 (strongly agree) to 4 (strongly disagree). The total raw score ranged from 7 to 28, with a higher score indicating a higher level of perceived mastery.
Achievement motives | about three months
  The Achievement Motives Scale (AMS) consists of two kinds of motives, referred to as Motive to Achieve Success, (MAS) and Motive to Avoid Failure (MAF). A short-form scale with 10 items was used to measure achievement motives, with 5 items each for MAS and MAF. Each item was scored on a Likert-type scale from 1 (strongly agree) to 4 (strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Long Guo, PhD, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan